CLINICAL TRIAL: NCT02182908
Title: ANALYSE EN MORPHO-TEP AU FDG DE L'EVOLUTIVITE DES ANEVRISMES ABDOMINAUX AORTIQUES NON CHIRURGICAUX UNE ETUDE MULTICENTRIQUE DE L'INTER-REGION NORD-EST
Brief Title: FDG PET-Scan Analysis of Evolutivity of Non-surgical Aneurysm of Abdominal Aorta
Acronym: AAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2006-004852-19
Record Dates: First submitted 2014-06-10; First posted 2014-07-08 (Estimated); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Medically-treated Aneurysm of Abdominal Aorta
Keywords: Aneurysm of abdominal aorta; 18F-fluorodesoxyglucose (FDG-F18)
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Non surgical aneurysm of abdominal aorta (Other): PET-Scan
  Interventions: Other: PET-Scan

INTERVENTIONS:
Other: PET-Scan — PET-Scan

SUMMARY:
The primary aim of the study is to determine if the evolutivity of global and segmentary captation of FDG-F18, which can be measured in the wall of abdominal aorta aneurysm, is predictive of the 9 month evolution of diameter and volume of the aneurysm, measured globally and segmentary in angioscan.

ELIGIBILITY:
Inclusion Criteria:

* AAA with a minimum diameter of 40 mm, calculated with a standardized method
* No indication for an immediate surgery or endoprothesis implantation
* Age above 18 (except for patient under supervision)
* Patient having read the information letter and signed the informed consent

Exclusion Criteria:

- AAA should have no other specific cause than atherosclerosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Association between overall baseline 18-FDG uptake intensity of the aneurysm and its 9-month maximal diameter and/or volume in patients with diameter change greater than 4 mm/year | 9 months
  Composite primary outcome.

SECONDARY OUTCOMES:
Association between initial 18-FDG uptake of individual aneurysmal segments and their 9-month diameter change. | 9 months
Contribution of overall 18-FDG uptake to the predictive values of other baseline characteristics of the aneurysm (diameter, volume, thickness and wall stress, clinical and biological values) | 9 months
Association between overall 18-FDG uptake and other baseline characteristics of the aneurysm (diameter, volume, thickness and wall stress, clinical and biological values). | 9 months
Association between 9-month overall 18-FDG uptake change and variation of plasmatic biomarkers of inflammation, proteolysis and coagulation. | 9 months

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Service de Médecine Nucléaire - CHU JEAN Minjoz, Besançon
  - CHU de Nancy - Hôpital Brabois, Vandœuvre-lès-Nancy